CLINICAL TRIAL: NCT04228900
Title: Nutrition and Medication Management in Home-dwelling Older Adults. Study II: Malnutrition in Older Adults: An Intervention Based on Medication Review and Individual Nutritional Plan
Brief Title: Malnutrition in Older Adults: An Intervention Based on Medication Review and Individual Nutritional Plan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Oslo (Other)
Collaborators: The Norwegian Research Fund for General Practice (Unknown)
Responsible Party: Principal Investigator, Mari Fiske, Principal investigator, University of Oslo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/12883-2
Record Dates: First submitted 2019-12-27; First posted 2020-01-14 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Malnutrition; Polypharmacy; Aged
Keywords: Malnutrition; Polypharmacy; Drug side effects; Nutritional improvement; Medication review
MeSH Terms: conditions — Malnutrition; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: A pragmatic clinical controlled study. Intervention in one municipality. Participants in neighbor municipality will comprise control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Drug review and tailored nutritional supply.
  Interventions: Dietary Supplement: Individualized plan for improvement of nutrition; Drug: Systematic drug review
- Control group (No Intervention): Follow-up by home nurse service and family physician "as usual".

INTERVENTIONS:
Dietary Supplement: Individualized plan for improvement of nutrition — For each participant we will make a plan, describing different items the can improve their nutritional status: enrichment of food, dental care,
  Arms: Intervention group
Drug: Systematic drug review — Consider altering medication list if the patient has symptoms that may be attributed to adverse drug effects, in particular side effects as nausea, dry mouth or loss of appetite, and if drug-drug interactions or drug-disease interactions are likely to occur. Recommended changes in patient's medication list will be presented for the family physician who will hold the final decision to implement the suggested adjustments.
  Arms: Intervention group

SUMMARY:
The project "Nutrition and Medication management in home-dwelling older adults" consist of two separate studies witch are described in the same study protocol. This is the second study in this Project. The first study (cross sectional) is described separately; Identification: 2017/12883-1

Undernutrition is common in older adults. The causes are many and include drug therapy. Drug side effects, as loss of appetite, nausea, or dry mouth, may contribute to malnutrition, impaired health and loss of function.

In patients with malnutrition or at risk for malnutrition we will evaluate an intervention consisting of:

* an "individual nutritional plan" with different measures aiming at improving nutritional status.
* a systematic drug review.

DETAILED DESCRIPTION:
The participants will be recruited by the home nursing services or by a nurse at a short-time ward in the nursing home.

The composite intervention consists has two components (A and B):

Component A: Clinical assessment and critical medication review

Drawing on information from the medical history, clinical finding according to examination made by the principal investigator (trained physician), information from the General Practitioner (GP) and the findings from blood tests, we will make a systematic and critical medication review. This systematic review has the following considerations:

* Are drug-drug unintended interactions likely to occur? Interaction analysis supported by https:// www.interaksjoner.no
* Are there use of potentially inappropriate medication? Assessed based on the Norwegian General Practice Nursing -Home criteria.
* Could nutritional related problems like loss of appetite, dry mouth and nausea, be attribute to adverse drug effects? Assessed by the list we made of drugs who often contributes to these side effects according to The Norwegian Pharmaceutical Product Compendium.

Component B: Nutritional intervention- individual nutrition plan. Drawing on the principles for good nutritional practice, and National guidelines, this component include the following considerations:

* Nutritional status by use of Mini Nutritional Assessment short form (MNA-SF), and further in- depth nutrition assessment if MNA-SF is in range 0-11.
* Assessment of the nutritional needs.
* Assess food and drink intake with a 3- day dietary record to the estimated nutritional needs.
* In collaboration with the home nurse, the participant and if possible/ necessary a next to kin, focusing on individual problems and develop an individual nutritional plan.

The project is about a controlled implementation of measures recommended in current national guidelines. We will follow a principle known as the "Nutritional Stairs", and choose interventions in the nutritional plan as close to "normal" food as possible. This means that the individual nutritional plan takes into account:

* Physical and mental disorders are diagnosed and optimal treated. (Oral health care included)
* Intervention to optimize the meal environment and meal itself, e.g., enough light in the room, specific tools to make eating possible if necessary, company
* The frequency of meals, length of night fasting, special diets as energy- and nutrient dens diets, consistency customized diet (liquid or solid food)
* Enriched food and in between meals/snacks
* Nutritional supplements

The intervention last six months, and participants in the intervention group will receive four visits at home; baseline and after 4, 12 and 24 weeks. At baseline and at week 24, the principal investigator (trained physician) and the nurse will visit the participants. At week 4 and 12, only the nurse will visit them. The control group, are visited by a nurse twice: at baseline and after 24 weeks, and are follow-up by the home nurse service and their GP "as usual".

Drop- out during the study period and reasons for "loss to follow-up (LTFU)" will be registered; e.g., moved from the municipality, acute illness that make further participation difficult, admission to long time ward in nursing home, or any other reason to withdraw participation. In the intervention group, we will on behalf of and subject to the participant's consent, make an appointment for consultation by the GP, if the clinical assessment suggests undetected diseases or diseases not optimal treated. If oral health problems are encountered, we will recommend a consultation by a dentist.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 year or more
* Receiving home nurse care each second week or more often
* Mini Nutritional Assessment short form (MNA-SF): 0-11 point (malnourished or at risk for malnutrition)

Exclusion Criteria:

* Life expectance less than 6 month
* Serious cognitive impairment
* In need of enteral-/ parenteral nutrition
* Not able to stand up for weight measure
* The home care service are not responsible for medication delivery.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-24 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Body weight at 24th week | Baseline, 24th week
  measurement of the participants weight

SECONDARY OUTCOMES:
Change from Baseline Health- related quality of life at 24th week | Baseline, 24th week
  answered by one question:"Consider your health, would you say it is: excellent(score 5)- very good (score 4)- good (score 3)- pretty good (score 2)- bad(score 1)" minimum score 1, Maximum score 5.The higher score the better.
Change from Baseline Activity of Daily living (ADL) at 24th week | Baseline, 24th week
  Assessed by Barthel´s ADL-index. Minimum score 0, Maximum score 20. The higher score the better.
Change from Baseline Admission to nursing home at 24th week | Baseline, 24th week
  Changes in Number of admissions to nursing home
Change from Baseline Admission to hospital at 24th week | Baseline, 24th week
  Change in Number of admissions to hospital
Change from Baseline Mini Nutritional Assessment short form (MNA-SF) at 24th week | Baseline, 24th week
  minimum score 0, Maximum score 14. 0-7 indicate malnutrition, 8-11 indicate risk for malnutrition, 12-14; normal nutritional status
Change from Baseline Number of drugs in daily use at 24th week | Baseline, 24th week
  Change in number of drugs in daily use
Change from Baseline Number of drugs in daily use considered inappropriate at 24th week | Baseline, 24th week
  Number of drugs considered inappropriate according to the Norwegian Practice Nursing-Home criteria, se protocol page 19-20,attachment 1
Change from Baseline Number of drugs in daily with high risk causing nausea, loss of appetite, and dry mouth at 24th week. | Baseline, 24th week
  See list Protocol page 21-23, attachment 2

CONTACTS AND LOCATIONS:
Overall Officials: Straand Jørund, Professor, Study Chair — Institute of Health and Society, University of Oslo, Norway
Locations (1):
- Department of General Practice, Institute og Health and Society, University og Oslo, Oslo, Norway

DOCUMENTS (5):
  • Informed Consent Form: participant, intervention group (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT04228900/ICF_000.pdf
  • Informed Consent Form: next of kin, intervention group (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT04228900/ICF_001.pdf
  • Informed Consent Form: participant, control group (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT04228900/ICF_002.pdf
  • Informed Consent Form: next of kin, control group (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT04228900/ICF_003.pdf
  • Study Protocol (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT04228900/Prot_004.pdf